CLINICAL TRIAL: NCT00807157
Title: Evaluation Des Effets Anti-Stress D'un Probiotique Nomme PROBIOSTICK® Sur Des Sujets Humains Volontaires Sains Sensibles Au Stress De La Vie Quotidienne
Brief Title: Evaluation of a Probiotic On Anxiety and Stress in Healthy Adults Sensible to Daily Stress
Acronym: BIOSTRESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Rosell Lallemand (Industry)
Responsible Party: Docteur Jean Marc Cazaubiel, Biofortis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BIOSTRESS 11008
Record Dates: First submitted 2008-12-08; First posted 2008-12-11 (Estimated); Last update posted 2009-04-24 (Estimated); Status verified 2009-04

CONDITIONS: Anxiety; Stress
Keywords: PROBIOSTICK®; Probiotic; Anxiety; Daily stress
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Placebo Comparator): Every morning subjects will consume a stick of placebo during 30 days
  Interventions: Dietary Supplement: Placebo during 30 days
- 1 (Experimental): Every morning subjects will consume a stick of PROBIOSTICK® during 30 days
  Interventions: Dietary Supplement: PROBIOSTICK® during 30 days

INTERVENTIONS:
Dietary Supplement: PROBIOSTICK® during 30 days — Every morning subjects will consume a stick of PROBIOSTICK® during 30 days
  Arms: 1
Dietary Supplement: Placebo during 30 days — Every morning subjects will consume a stick of placebo during 30 days
  Arms: 2

SUMMARY:
The purpose of the the study is to determine if PROBIOSTICK® decrease stress and anxiety of people sensible to daily stress.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian healthy men or women
* Age 30-60 years
* Hospital anxiety and depression score equal or below 12 and above 4
* Standard safety biology

Exclusion Criteria:

* HAD A results above 12 and below 4
* HAD D results above 12
* Neurologic or psychiatric pathology
* Consumption of psychotropic
* High level of caffeine consumption
* Any important chronic pathology
* Drugs wich impairs concentration, anxiety and stress

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
SCL 90 questionnaire | day 0 and day 30

SECONDARY OUTCOMES:
Stress perçu, coping de vitaliano, hospital anxiety and depression questionnaires and urinary cortisol measurement | day-14 ; day 0 and day 30

CONTACTS AND LOCATIONS:
Locations (1):
- Biofortis, Nantes, France